CLINICAL TRIAL: NCT05451524
Title: Prevention of Insomnia in At-risk Youth: A Randomized Controlled Trial Comparing Cognitive Behavioural Prevention Programme for Insomnia With Active Control Condition
Brief Title: Prevention of Insomnia in At-risk Youth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHAN NGAN YIN, Research Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021.005
Record Dates: First submitted 2022-06-18; First posted 2022-07-11 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Insomnia
Keywords: insomnia; prevention; at-risk youth; cognitive behavioral approach; active control group
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Assessors and statisticians, participants will be masked to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insomnia prevention program (Experimental): The preventive program has been developed and modified as based on the evidence-based CBT-I insomnia treatment.
  Active intervention group will be conducted in group size with 6-8 subjects who are from the same education level (i.e. secondary vs university). Youths in the intervention group will receive 4 weekly insomnia prevention program conducted by the sleep therapists who has received training in conducting CBT-I under close supervision of sleep experts. Each session will last for about 60-90 mins.
  Interventions: Behavioral: Insomnia prevention program
- General health education (Active Comparator): In order to control for placebo effect and other non-specific factors such as contact time, youths in the control group will be provided with group-based general health education with same dosage (4 weeks) as intervention group. Modules will contain information about general well-being, diet, nutrition, and activity. It is expected that this health education will be an active control group to account for most of the non-specific effects including time, attention, therapist, and peer support.
  Interventions: Behavioral: General health education

INTERVENTIONS:
Behavioral: Insomnia prevention program — Youths in the intervention group will receive 4 weekly insomnia prevention program. Each session will last for about 60-90 mins.
  Arms: Insomnia prevention program
Behavioral: General health education — Youths in the control group will be provided with group-based general health education with same dosage (4 weeks) as intervention group.
  Arms: General health education

SUMMARY:
This study aims to conduct a randomized controlled trial in comparing cognitive behavioral insomnia prevention program with the active control group in youths who are at risk of insomnia. The results of this study will allow us to take this potential efficacious prevention program to scale and reduce the associated burden of insomnia in the future.

DETAILED DESCRIPTION:
Adolescence is a vulnerable period for the emergence of insomnia, which affects more than 10% of the youths (approximately 40% if based on symptoms). Insomnia in youths tends to run a protracted course and is associated with numerous negative outcomes including poor quality of life, cognitive and academic impairment, and predisposing to development of depression and anxiety. The burden arises from insomnia has been increasingly recognized worldwide as a debilitating and costly public health concern.

However, insomnia in youths is often ignored and under-treated, with only 10% of the local youths recognized their insomnia problem and none of them has received the recommended first-line treatment - cognitive behavioral therapy for insomnia (CBT-I). Given the high prevalence, chronicity and long-lasting health-related consequences of insomnia, together with the delay and limited help-seeking behavior, it calls the urgent need for early insomnia prevention and intervention in this vulnerable population.

Thus, this study aims to conduct a randomized controlled trial in comparing cognitive behavioral insomnia prevention program with the active control group in youths who are at risk of insomnia and to explore the effect of prevention program in preventing the incidence of insomnia problems.

ELIGIBILITY:
Inclusion Criteria:

* Youth aged between 15-24 years (as defined by WHO);
* Written informed consent of participation into the study is given by youth and his/her parents if under 18 years old; In addition, individual assent will also be obtained for subjects under age 18 years old;
* Have subclinical insomnia symptoms (at least once a month but less than 3 times/week in the past one month);
* At least one of the biological parents with current or lifetime history of insomnia disorder as defined by DSM-V diagnostic criteria.

Exclusion Criteria:

* A current or past history of neuropsychiatric disorder(s);
* A prominent medical condition or taking medication with potential side effects that may influence sleep quantity and quality;
* Having a diagnosed sleep disorder that may potentially contribute to the disruption of sleep quantity and quality as ascertained by both Structured Diagnostic Interview for Sleep patterns and Disorders (DISP) such as insomnia, delayed sleep phase and narcolepsy, restless leg syndrome;
* Having a clinically significant suicidality (presence of suicidal ideation with a plan or an attempt);
* Currently receiving any structured psychotherapy;
* With hearing or speech deficit;
* Trans-meridian flight in the past 3 months and during the study.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 204 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Insomnia disorder incidence | week 5
  Clinician-rated insomnia incidence is defined as having insomnia symptoms for ≥ 3 times per week for at least one month (will be able to cover both acute and chronic insomnia disorder), accompanied with clinically significant distress or impairment. The assessment will be conducted based on the DSM-V insomnia diagnostic criteria checklist with the detail record of the symptom duration.
Insomnia disorder incidence | 3-month follow up
  Clinician-rated insomnia incidence is defined as having insomnia symptoms for ≥ 3 times per week for at least one month (will be able to cover both acute and chronic insomnia disorder), accompanied with clinically significant distress or impairment. The assessment will be conducted based on the DSM-V insomnia diagnostic criteria checklist with the detail record of the symptom duration.
Insomnia disorder incidence | 6-month follow up
  Clinician-rated insomnia incidence is defined as having insomnia symptoms for ≥ 3 times per week for at least one month (will be able to cover both acute and chronic insomnia disorder), accompanied with clinically significant distress or impairment. The assessment will be conducted based on the DSM-V insomnia diagnostic criteria checklist with the detail record of the symptom duration.
Insomnia disorder incidence | 12-month follow up
  Clinician-rated insomnia incidence is defined as having insomnia symptoms for ≥ 3 times per week for at least one month (will be able to cover both acute and chronic insomnia disorder), accompanied with clinically significant distress or impairment. The assessment will be conducted based on the DSM-V insomnia diagnostic criteria checklist with the detail record of the symptom duration.
Change of insomnia symptoms | baseline, week 5, 3-, 6-, and 12-month follow up
  The severity of insomnia symptoms as measured by 7-item Insomnia Severity Index (ISI). ISI is a self-report measure designed to assess the nature, severity and impact of insomnia, with a higher total score suggesting more severe insomnia symptoms. Scores range from 0 to 28.

SECONDARY OUTCOMES:
Change of sleep parameters as measured by 7-day sleep diary | baseline, week 5, 3-, 6-, and 12-month follow up
  Seven-day sleep diary is a prospective measure that includes the questions to assess time in bed, sleep duration, wake after sleep onset, sleep latency and sleep efficiency.
Change of score in vulnerability to stress-related insomnia | baseline, week 5, 3-, 6-, and 12-month follow up
  Vulnerability to stress-related insomnia will be measured by Ford Insomnia Response to Stress Test (FIRST). It includes nine items, and participants were asked to rate on a 4-point Likert scale to indicate their likelihood of sleep disturbance in response to the commonly experienced stressful situations. A higher total score represents a greater vulnerability of sleep disturbance. The total score ranges from 9 to 36.
Change of sleep-related thoughts and behaviors | baseline, week 5, 3-, 6-, and 12-month follow up
  Sleep-related thoughts and behaviors will be measured by Brief Version of Dysfunctional Beliefs and Attitudes about Sleep (DBAS-16). DBAS-16 is a 16-item self-report measure designed to evaluate a subset of those sleep related cognition, with a higher score indicating more dysfunctional beliefs and attitudes about sleep. The total score is calculated from the average score of all the items on the scale and could range from 0 to 10.
Change of daytime sleepiness | baseline, week 5 3-, 6-, and 12-month follow up
  Daytime sleepiness will be measured by Pediatric Daytime Sleepiness Scale (PDSS). It is an 8-item inventory designed for use with school children and youths, with a higher score indicating greater sleepiness. Scores ranged from 0 to 32.
Daytime fatigue | baseline, week 5, 3-, 6-, and 12-month follow up
  Daytime fatigue will be assessed by Multidimensional Fatigue Inventory (MFI) that measure five dimensions of fatigue, including general fatigue, physical fatigue, mental fatigue, reduced motivation and reduced activity. MFI is a self-report instrument consisting of 20 items. Each subscale contains four items. The total scores of each subscale range from 4 to 20, with a higher score indicating greater fatigue.
Change of self-reported cognitive failures | baseline, week 5, 3-, 6-, and 12-month follow up
  Cognitive Failures Questionnaire (CFQ) is an indicator of self-reported failures in perception, memory, and motor function, with a higher score indicating an increased vulnerability to stress. Scores range from 0 to 100.
Change of anxiety and depressive symptoms | baseline, week 5, 3-, 6-, and 12-month follow up
  Anxiety and depressive symptoms will be measured by Hospital Anxiety and Depression Scale (HADS). The HADS consists of two subscales for anxiety (HADS-A) and depression (HADS-D). A higher total score of each subscale represents a greater severity of depression/anxiety. The total score for each subscale ranges from 0 to 21.
Change of health related quality of life | baseline, week 5, 3-, 6-, and 12-month follow up
  Quality of life will be measured by kidscreen-27 Health related quality of life (HRQoL) that consists of 27 items to assess five dimensions of quality of life, including physical well-being (possibly scored from 5 to 25), psychological well-being (possibly scored 7 to 35), autonomy & parents (possibly scored 7 to 35), peers & social support (possibly scored 4 to 20), and school environment (possibly scored 4 to 20). A grand total score can be calculated by summing up the five sub scores. In all cases, a higher score represents higher perceived well-being.
Change of sleep hygiene | baseline, week 5, 3-, 6-, and 12-month follow up
  Adolescent sleep behaviors will be measured by Adolescent Sleep Hygiene Scale revised (ASHSr). ASHSr is a self-reported questionnaire with eight subscales: physiological, cognitive, emotional, sleep environment, daytime sleep, substance, sleep stability and bedtime routine. A higher score indicates a better sleep practice. The total score is calculated from the average score of all the items on the scale and could range from 1 to 6.
Change of pre-sleep arousal behaviors | baseline, week 5, 3-, 6-, and 12-month follow up
  Pre-Sleep Arousal Scale (PSAS) is a 16-item, self-reported questionnaire comprising both cognitive and somatic manifestations of arousal, with eight items in each subscale. Two subscale scores ranging from 8 to 40 were computed separately. A higher score suggesting higher pre-sleep arousal.
Change of academic performance | baseline and 12-month follow up
  Official record of academic performance at both baseline and end of study (at 12 months) will be collected.
Change of adolescent's perception and attitude towards sleep | baseline, week 5 3-, 6-, and 12-month follow up
  Adolescent's perception and attitude towards sleep will be captured by 10-item Charlotte Attitudes Towards Sleep Scale (CATS). The CATS Scale included 2 subscales: the Benefits subscale the Time Commitment subscale. The 5 items within each subscale can be averaged, and all 10 items can be averaged to create a total score ranging from 1 to 7, with higher scores indicating more favorable attitudes towards sleep.

OTHER OUTCOMES:
Major life events and self-perceived stress | baseline and 12-month follow up
  Major life events and self-perceived stress associated with these events that an individual experienced over the year will be measured by 57-item Life Experience Survey (LES). Ratings are on a 7-point scale ranging from extremely negative (-3) to extremely positive (+3). Summing the impact ratings of those events designated as positive by the subject provides a positive change score. A negative change score is derived by summing the impact ratings of those events experienced as negative by the subject. By adding these two values, a total change score can be obtained, representing the total amount of rated change, and can range from 0 to 171.
Change of chronotype | baseline, week 5, 3-, 6-, and 12-month follow up
  The chronotype of the study participants will be measured by Morningness-Eveningness Questionnaire (MEQ). The rMEQ is a 5-item self reported measure used to evaluate circadian rhythm and sleep rhythm patterns in individuals. Individuals scored higher than 17 and lower than 12 were classified as morning-type and evening-type, respectively. Individuals scored between 12 and 17 were classified as intermediate-type. Scores range from 4 to 25.
Self-reported pubertal status | baseline and 12-month follow up
  Tanner staging of breasts for females or genitals for males and pubic hair presented in pictures with text descriptions will be used to determine the pubertal status. A rating falls between tanner stages of one to three is classified as the pre-pubertal stage, while tanner stages four and five is classified as the post-pubertal stage.
Treatment satisfaction, adherence and integrity | week 5
  The TSS consists of 7 items with higher scores indicating greater symptom improvement. Overall treatment satisfaction was computed as the average score which ranges from 1 to 5 on all 7 items of the TSS.
Treatment adherence | week 5
  Treatment Component Adherence Scale (TCAS) will be used to assess treatment adherence at post intervention. The TCAS consists of 6 items with higher scores indicating better adherence. Scores range from 0 to 18
Treatment expectancy and credibility | week 5
  Credibility-Expectancy Questionnaire (CEQ) for assessment of treatment expectancy and credibility of the intervention. The CEQ consists of 6 items with higher scores indicating greater perceptions of treatment credibility and expectations of improvement. Scores range from 5 to 30.

CONTACTS AND LOCATIONS:
Overall Officials: NGAN YIN CHAN, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Psychiatry, Shatin, NT, Hong Kong

IPD SHARING:
Plan to Share IPD: No